CLINICAL TRIAL: NCT06006832
Title: Clinical Characteristics, Prognosis and Biomarkers of Myasthenia Gravis: a Prospective Cohort Study in China
Brief Title: A Prospective Cohort Study of Myasthenia Gravis in China
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K2009
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-08

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood of each participant at each visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- maintenance steroid therapy group: Maintaining low-dose oral steroids
  Interventions: Drug: Steroid Drug
- immunosuppresants withdrawal group: Withdraw all immunosuppresants
  Interventions: Other: Withdraw all immunosuppresants

INTERVENTIONS:
Drug: Steroid Drug — Maintaining low-dose oral steroids
  Groups: maintenance steroid therapy group
Other: Withdraw all immunosuppresants — Withdraw all immunosuppresants
  Groups: immunosuppresants withdrawal group

SUMMARY:
The goal of this prospective cohort study is to investigate long-term therapeutic strategies for myasthenia gravis (MG) and identify potential biomarkers. The main questions it aims to answer are:

1. Whether low-dose oral steroids may lead to a reduction in the recurrence rate among patients with MG.
2. To identify potential biomarkers that can predict disease progression and prognosis.

This study recruits well-controlled patients with MG. Based on patient preferences and considerations such as coexisting conditions (e.g., uncontrolled hypertension, diabetes, severe osteoporosis, obesity), the participants will be non-randomly divided into two groups: a maintenance steroid therapy group and a withdrawal group (withdraw all immunosuppresants). Subsequently, these groups of patients will undergo long-term follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* 1: Attended the outpatient department of neurology of PUMCH from 9/30/2022 to 9/30/2024.
* 2: Diagnosed as myasthenia gravis.
* 3: Follow-up time at PUMCH>6 months.
* 4: The patient understood and signed the informed consent form.

Exclusion Criteria:

* 1: Comorbidities with other conditions that cause skeletal muscle weakness make the clinical symptoms difficult to assess
* 2: Records related to comorbidities and medications were not available at baseline and during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myasthenia gravis who can completed long-term follow-up at PUMCH.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Relapse of myasthenia gravis | Within two years after recruitment
  One of the following three is met: (1) MGFA Postintervention Status: failure to maintain MMS (minimal manifestations status) or better. (2) Myasthenia gravis activities of daily living (MG-ADL) score ≥ 3; (3) Re-administration of cholinesterase inhibitors was required after achieving Complete Stable Remission (CSR) on the MGFA Postintervention Status.

SECONDARY OUTCOMES:
Time of relapse | Within two years after recruitment
  The time between recruitment and relapse of MG.
Change of MG assessment scales at relapse | Within two years after recruitment
  Change of MG assessment scales at relapse, including MGFA PIS (Postintervention Status), MG-ADL (myasthenia gravis activities of daily living), QMG (Quantitative Myasthenia gravis) and MGC (Myasthenia gravis composite).
Adverse events of steroids | Within two years after recruitment
  Using CTCAE (Common Terminology Criteria for Adverse Events) to assess Adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yuzhou Guan, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No